CLINICAL TRIAL: NCT03192371
Title: A Phase IV, Randomized, Open-label Study to Evaluate One Year Long-term Persistence of Immune Responses Following Two Different Rabies Vaccine Post-exposure Regimens (Zagreb 2-1-1 and Essen 1-1-1-1-1) in Chinese Children
Brief Title: A Study to Evaluate the One Year Long-term Persistence of Immune Responses Following Two Different Rabies Vaccine Post-exposure Regimens in Chinese Children
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to supply constraints & prioritization according to medical need (availability of alternative rabies vaccines), Rabipur will no longer be supplied to China.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205854
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Virus Diseases
Keywords: Zagreb regimen; Encephalitis; Antibody persistence; Essen regimen; Post-Exposure Prophylaxis (PEP); Rabies
MeSH Terms: conditions — Virus Diseases; Encephalitis; Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects will be stratified into age subsets of equal numbers within each age cohort (children: 6 to11 years of age and 12 to 17 years of age). Within each age subset, subjects will be assigned randomly in a 1:1 ratio, to one of the two regimens: Zagreb (2-1-1) Group and Essen (1-1-1-1-1) Group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zagreb 2-1-1 Group (Experimental): 4 doses of Rabipur vaccine, administered intramuscularly according to the Zagreb (2-1-1) regimen (i.e., 2 doses of vaccine administered on Day 1 and 1 dose of vaccine administered on Days 8 and 22).
  Interventions: Biological: Rabipur
- Essen 1-1-1-1-1 Group (Experimental): 5 doses of Rabipur vaccine, administered intramuscularly according to the Essen (1-1-1-1-1) regimen (i.e., 1 dose of vaccine administered on Days 1, 4, 8, 15, and 29).
  Interventions: Biological: Rabipur

INTERVENTIONS:
Biological: Rabipur — Rabies vaccine administered as an intramuscular injection according to Zagreb or Essen regimen to subjects aged ≥6 to ≤17 years.
  Other Names: Rabies Vaccine (Chicken Embryo Cell) for Human use

SUMMARY:
The purpose of this study is to evaluate the 1 year immunogenicity persistence of Rabipur in children 6-17 years of age, and compare the Zagreb regimen with the Essen regimen.

DETAILED DESCRIPTION:
The clinical basis for the last renewal of the Rabipur license in China was the results from study V49_24 (NCT01680016), an immunogenicity and safety trial conducted in Chinese children (6 to 17 years) and adults (≥51 years), which confirmed the non-inferior immunogenicity of the Zagreb versus the conventional Essen post exposure prophylaxis intramuscular (PEP IM) regimen at Day 15 for both age groups.

At the time of license renewal in 2015, the Chinese health authorities requested that GSK continue to conduct immunogenicity persistence follow-ups for at least 1 year to compare the Zagreb regimen with the Essen regimen in populations under 17 years old.

V49_24E1 is an extension study to meet this request, in which subjects aged 17 years or younger who were immunized in the parent trial V49_24 will be recalled for a blood immunogenicity analysis approximately 4-5 years after the original vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of 6 through 17 years of age on the day of informed consent/assent.
2. Individuals who are in good health at the time of entry into the study as determined by medical history, physical examination and clinical judgment of the investigator.
3. Individuals who or whose parent(s)/legal guardian(s) have voluntarily given written informed consent on behalf of their child, and adolescents who have provided written assent, after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
4. Individuals who can comply with study procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. A body temperature ≥38°C (axillary) within 3 days of intended study vaccination.
2. Known hypersensitivity to gentamycin, known allergies to excipients of Rabipur such as Polygeline, chicken protein, egg products or any other vaccine component.
3. Previously received any rabies vaccine or rabies immune globulin.
4. Subjects currently receiving or planning to receive antimalarial medications 4 days prior to V1/Day 1 vaccination and until the final vaccination.
5. Progressive, unstable or uncontrolled clinical conditions.
6. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
7. Abnormal function of the immune system resulting from:

   1. Clinical conditions.
   2. Systemic administration of corticosteroids for more than 14 consecutive days within 90 days prior to informed consent.
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
8. Received immunoglobulins or any blood products within 180 days prior to informed consent.
9. Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
10. Study personnel as an immediate family or household member.
11. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.
12. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.
13. Children in care: A child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a child in care can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or has an appointed legal guardian.
14. If female of childbearing potential and sexually active, refusal to use an "acceptable contraceptive method" for the duration of the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2019-05-12 (Estimated); Study Completion 2019-05-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of immunogenicity in terms of antibody concentrations. | Study days 1, 15, 43, 197 and 393.
  Immunogenicity is assessed in terms of Geometric Mean Concentration (GMC) of Rabies Virus Neutralizing Antibody (RVNA) concentrations.
  Comparison between Zagreb and Essen groups will be reported in terms of difference between GMCs.
Percentage of subjects with RVNA concentrations ≥ 0.5 IU/mL | Study days 1, 15, 43, 197 and 393.
  Comparison between Zagreb and Essen groups will be reported in terms of difference between percentages of subjects with RVNA concentrations ≥ 0.5 IU/mL.
All Serious Adverse Events (SAEs) and Adverse Events (AEs) leading to subject withdrawal. | From Day1/Visit 1 through Day 393/Visit 11 (study termination).
  Only SAEs and unsolicited AEs leading to study withdrawal will be collected. SAEs to be assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of existing hospitalization, result in disability/incapacity, result in congenital anomaly/or birth defect or significant medical event that may not be immediately life threatening or resulting in death or hospitalization but may jeopardize the subject or require intervention to prevent one of the other outcomes listed.
  An unsolicited AE is an AE that was not solicited using a Subject Diary and that was spontaneously communicated by a subject and/or parent(s)/legal guardian(s) who has signed the informed consent. Potential unsolicited AEs may be medically attended (defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider), or were of concern to the subject and/or parent(s)/legal guardian(s).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: No